CLINICAL TRIAL: NCT06111872
Title: Combination Use of Intravenous Ketamine-midazolam as a Sedative Agent in Endoscopic Retrograde Cholangiopancreatography ; A Randomized Control Trial
Brief Title: Ketamine-midazolam as a Sedative Agent in Endoscopic Retrograde Cholangiopancreatography.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Prof Madya Dr. Azlanudin Azman, Associate Professor, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JEP-2023-272
Record Dates: First submitted 2023-10-12; First posted 2023-11-01 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-10

CONDITIONS: Cholangitis; Pancreatic Cancer; Choledocholithiasis; Choledochal Cyst
Keywords: Ketamine; Midazolam; sedation; ERCP
MeSH Terms: conditions — Cholangitis; Pancreatic Neoplasms; Choledocholithiasis; Choledochal Cyst | interventions — Ketamine; Midazolam; Meperidine

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into the intervention or control group (Intervention group will receive Ketamine - Midazolam and control group will receive Midazolam- Pethidine as a sedative agent in ERCP
Who Masked: Care Provider
Masking Description: Care provider is blinded from knowing the group of the study. However patients are informed regarding the drugs received
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine - Midazolam arm (Experimental): Initial IV Ketamine of 0.5mg/kg with IV Midazolam 0.02mg/kg given over 1 minute. If depth of sedation not adequate, to give another bolus of IV ketamine 0.25mg/kg after 2 minutes with IV Midazolam 0.01mg/kg. If depth of sedation not adequate, to give another bolus of IV Ketamine 0.25mg/kg after 2 minutes and IV Midazolam 0.01mg/kg. Failure of sedation: inadequate sedation for the intention to treat: patient will be arranged for MAC (monitored anaesthesia care) with anaesthesia team
  Interventions: Drug: Ketamine; Drug: Midazolam
- Midazolam - Pethidine arm (Active Comparator): Initial IV Midazolam 0.05mg/kg given over 1 minute with IV Pethidine 0.7mcg/kg. If depth of sedation not If adequate, to give another bolus of IV Midazolam 0.02mg/kg after 2 minutes and IV Pethidine 0.7mcg/kg. If depth of sedation not adequate, to give another bolus of IV Midazolam 0.02mg/kg after 2 minutes. Failure of sedation: inadequate sedation for the intention to treat: patient will be arranged for MAC (monitored anaesthesia care) with anaesthesia team.
  Interventions: Drug: Midazolam; Drug: Pethidin

INTERVENTIONS:
Drug: Ketamine — Administration described in arm/ group description
  Other Names: KETAMINE- MIDAZOLAM
  Arms: Ketamine - Midazolam arm
Drug: Midazolam — Administration described in arm/ group description
  Other Names: KETAMINE-MIDAZOLAM
Drug: Pethidin — Administration described in arm/ group description
  Other Names: MIDAZOLAM-PETHIDIN
  Arms: Midazolam - Pethidine arm

SUMMARY:
Does Ketamine-Midazolam have a better efficacy and safety profile compared to Midazolam - Pethidine in Endoscopic Retrograde Cholangiopancreatography (ERCP)?

DETAILED DESCRIPTION:
Ketamine- Midazolom is more efficacious in producing desired sedative state and have a better safety profile as a sedative agent in ERCP compared to Midazolam- Pethidine. The usage of sedative agent in ERCP depends on surgeon's preferences and availability of the drugs. The most commonly used sedatives in ERCP is Midazolam with pethidine. The use of Midazolam , however, is related to:

1. 20-45% failure of sedation during ERCP
2. Cardio-respiratory depression - apnoea: 15.4%, hypotension: 15.7%, bradycardia: 6.8%

Due to the proven efficacy and safety profile of ketamine-midazolam as a sedative agent in procedural sedation, the investigators propose that the use of ketamine-midazolam as a sedative agent in ERCP is more effective and better safety profile when compared to Midazolam- Pethidine. The synergistic effect means to reduce the total dose of midazolam used.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years old which able to give valid consent
* Patient planned for ERCP (either emergency or elective)
* American Society of Anaesthesiologist (ASA) score of I-III

Exclusion Criteria:

* Known hypersensitivity towards Ketamine or Midazolam
* Increased intracranial pressure, acute stroke (<3 months), intracranial haemorrhage (<3 months)
* Severe hypertension (BP>170/110) and tachycardia (Heart rate >110)
* Acute myocardial infarction, acute coronary syndrome (< 6 months)
* Tachyarrhythmia
* Pregnancy
* Intravenous drug user (IVDU) or substance abuse patient
* History of hallucination
* Child's Pugh class C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
To compare the depth of sedation | Evaluated at specific timepoints during the procedure whch are: introduction of scope, canulation of bile duct, trawling of stones, removal of stent and removal of scope
  The depth of sedation is evaluated using ramsay sedation scale where the scale is 1 to 6, where higher score is better

SECONDARY OUTCOMES:
To evaluate the efficacy of Ketamine- Midazolam as a sedative agent in ERCP in terms of sedation failure rate. | Evaluated at specific timepoints during the procedure whch are: introduction of scope, canulation of bile duct, during sphincerotomy, removal of stent and removal of scope
  Sedation failure rate is defined as inability of the sedation used to adequately sedate a patient for initiation and completion using ramsay sedation scale where the scale is 1-6, where higher score is better.
To compare pre and post procedure mean arterial pressure (MAP) | Measured at specific time-pointswhich are: pre-sedation, 2 minutes after initiation of sedation and 5 minutes after the procedure is completed
  To detect if there are changes in MAP calculated from participants blood pressure readings
To compare surgeon satisfaction in terms of sedation quality between both arms using a likert scale of 1 to 5 where a higher score is better | Single point asessment at the end of the procedure
  Measured using likert scale
To compare participant satisfaction in terms of procedure experience between both groups using likert scale of 1 to 10 where the higher score is better | Single point asessment at 2 hours after completion of procedure
  Measured using likert scale
To compare the number of participants that developed an adverse event that led to abandonment of procedure | Evaluated at specific timepoints during the procedure which are: introduction of scope, canulation of bile duct, during sphincerotomy, trawling of stones, removal of stent and removal of scope
  Adverse event by monitoring patient vital signs including blood pressure, pulse rate, oxygen saturation and procedure will be abandoned if the parameters reach a pre-set cut-off point.
  Systolic blood pressure <90mmHg or >180mmHg, Pulse rate of <60/min or >150/min and oxygen saturation <95% despite supplemental oxygen therapy via nasal canula.

CONTACTS AND LOCATIONS:
Overall Officials: Azlanudin Azman, Principal Investigator — Universiti Kebangsaan Malaysia Medical Centre
Locations (1):
- Hospital Canselor Tuanku Muhriz UKM, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
Currently undecided

REFERENCES:
- [Background] Narayanan S, Shannon A, Nandalan S, Jaitly V, Greer S. Alternative sedation for the higher risk endoscopy: a randomized controlled trial of ketamine use in endoscopic retrograde cholangiopancreatography. Scand J Gastroenterol. 2015;50(10):1293-303. doi: 10.3109/00365521.2015.1036113. Epub 2015 Jun 10. PMID 26061267
- [Background] Tobias JD, Leder M. Procedural sedation: A review of sedative agents, monitoring, and management of complications. Saudi J Anaesth. 2011 Oct;5(4):395-410. doi: 10.4103/1658-354X.87270. PMID 22144928
- [Background] Jung M, Hofmann C, Kiesslich R, Brackertz A. Improved sedation in diagnostic and therapeutic ERCP: propofol is an alternative to midazolam. Endoscopy. 2000 Mar;32(3):233-8. doi: 10.1055/s-2000-96. PMID 10718389
- [Background] Tokmak S, Cetin MF, Torun S. Efficacy and safety of endoscopic retrograde cholangiopancreatography in the very elderly by using a combination of intravenous midazolam, ketamine and pethidine. Geriatr Gerontol Int. 2021 Oct;21(10):887-892. doi: 10.1111/ggi.14252. Epub 2021 Aug 23. PMID 34427037
- [Background] Goudra B, Nuzat A, Singh PM, Borle A, Carlin A, Gouda G. Association between Type of Sedation and the Adverse Events Associated with Gastrointestinal Endoscopy: An Analysis of 5 Years' Data from a Tertiary Center in the USA. Clin Endosc. 2017 Mar;50(2):161-169. doi: 10.5946/ce.2016.019. Epub 2016 Apr 29. PMID 27126387